CLINICAL TRIAL: NCT03979274
Title: Prospective, Single Dose, Randomized, Open Label, Comparative, Cross-study to Establish Bioequivalence Between the New Formulation and the Approved Formulation for Levothyroxine (Eutirox® From Merck, S. A. de C. V.) Given as 3 Tablets of 200 μg p.o. in Healthy Volunteers
Brief Title: A Comparative Study of New Formulation and Approved Formulation for Levothyroxine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200125_0008
Record Dates: First submitted 2019-06-06; First posted 2019-06-07 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Eutirox; Levothyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference Eutirox®, then Test Eutirox® (Experimental): Participants received single oral dose of Reference Eutirox® 600 microgram (mcg) (3 tablets of 200 mcg) in Treatment Period 1 followed by single oral dosing of Test Eutirox® 600 mcg (3 tablets of 200 mcg) in Treatment Period 2. A wash-out period of 35 days was maintained between the Treatment Periods 1 and 2.
  Interventions: Drug: Reference Eutirox®; Drug: Test Eutirox®
- Test Eutirox®, then Reference Eutirox® (Experimental): Participants received single oral dose of Test Eutirox® 600 mcg (3 tablets of 200 mcg) in Treatment Period 1 followed by single oral dosing of Reference Eutirox® 600 mcg (3 tablets of 200 mcg) in Treatment Period 2. A wash-out period of 35 days was maintained between the Treatment Periods 1 and 2.
  Interventions: Drug: Reference Eutirox®; Drug: Test Eutirox®

INTERVENTIONS:
Drug: Reference Eutirox® — Participants received single oral dose of Reference Eutirox® 600 microgram (3 tablets of 200 microgram) either in treatment period 1 or 2.
Drug: Test Eutirox® — Participants received single oral dose of Test Eutirox® 600 microgram (3 tablets of 200 microgram) either in treatment 1 or 2.

SUMMARY:
The study investigated the bioequivalence between the new and the approved formulation for levothyroxine.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided their written consent prior to any study-related activity
* Ethnic origin: Mexicans
* Body mass index from 18 to 27 kilogram per meter square (kg/m^2)
* Normal vital signs (includes heart rate between 50 and 100 beats per minute, respiratory rate between 12 and 20 per minute, systolic blood pressure between 80 and 129 milimeter of mercury (mmHg) , diastolic blood pressure between 50 and 80 mmHg and temperature between 36.0 degree celsius and 37.0 degree celsius. The measurement will be made according to the instructive BE-IT-005 Medición de signos vitales)
* Normal electrocardiogram [ECG]. No abnormalities are allowed, even though they are not relevant (PR, QRS, QT, QTcF should be within normal range; no conduction abnormalities are allowed, etcetera (etc)
* All values in blood and urine tests should be within the normal range or showing no clinically relevant deviation as judged by the Investigator
* Participants with thyroid panel results within normal range (T3 and T4 total and free, as well as thyroid-stimulating hormone (TSH) should be within the normal range)
* Non-smoker at least in the last 3 months
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participation in the clinical study within 90 days prior to the first dose of the study drug
* History of hypersensitivity to the study drug or its excipients
* History or current asthma or any severe allergy (which requires hospitalization or prolonged therapy), allergy or intolerance to any food that, in the opinion of the investigator, poses a safety risk (allergy to iodine)
* History of cardiovascular, renal, liver, metabolic, gastrointestinal, neurological, endocrine, hematopoietic (any type of anemia) conditions, mental disorder or organic abnormalities that may affect the pharmacokinetic study of the study drug
* Any medical or surgical condition, including findings in the medical history or clinical assessment prior to the study, that in the opinion of the investigator poses a risk or contraindication for the participants participation in the study and may affect the study objectives, conduct or analysis
* History or presence of alcohol abuse (average daily intake not higher than 3 units or weekly intake not higher than 21 units; 1 unit is equivalent to 340 mililiter (mL) of beer, 115 mL of wine or 43 mL of prepared drinks), psychoactive substances or chronic use of drugs
* Participants who have been exposed to agents knows by inducing or inhibiting the liver enzymatic systems or who have taken potentially toxic drugs within the last 30 days to the study start-up
* Participants who take drugs affecting the metabolism of the thyroid hormone, such as: oral contraceptives, hormonal implants, parenteral hormones, steroids, anabolic drugs, androgens, etc., or any drug affecting the levothyroxine's bioavailability such as the proton pump inhibitors or multivitamins, nutritional supplements or herbal products that may affect the study, except for the occasional use of paracetamol
* Participants who have been hospitalized for any reason within the 60 days prior to the study start-up or who have been severely ill within the last 30 days prior to the study start-up
* Participants who have donated or lost 450 mL of blood within the last 60 days prior to the study start-up
* Participants non- smokers, who have smoked tobacco, cigarettes or consumed coffee, snuff or drinks containing xanthines such as caffeine, (tea, cocoa, chocolate, matte, cola, etc.) theobromine, theophylline, among others, affecting the pharmacokinetics of the drug in assessment, drinking alcohol, or charcoal-grilled foods consumed within twenty-four hours prior to administration the dose of medication
* Screening biosafety positive tests for the human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) and syphilis Venereal Disease Research Laboratory (VDRL)
* Positive result in the abuse drugs screening tests, such as: amphetamines, benzodiazepines, cocaine, methamphetamines, morphine and tetrahydrocannabinoids
* Presence of alcohol in breath test
* Women pregnancy positive tests (qualitative and quantitative) at the screening and inclusion in each period
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Cecype, Fray Bernardino de Sahagún, Morelia - Michoacan, Mexico

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany, will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — http://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200125_0008
- See also: Medical Information Location Map - Med Info Contacts — http://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Reference Eutirox®, Then Test Eutirox® | Test Eutirox®, Then Reference Eutirox®
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Reference Eutirox®, Then Test Eutirox® | Test Eutirox®, Then Reference Eutirox®
Started | 22 | 22
Completed | 22 | 21
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least one dose of study medication.
Groups:
- All Participants: All participants who received a single oral dose of Reference Eutirox® 600 mcg (200*3 mcg) or a single oral dose of test Eutirox® 600 mcg (200*3 mcg) in either Treatment Period 1 or 2.
Arm/Group | All Participants
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.93 (5.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration in Pre Dose Corrected Data (Cmax[aj]) of Levothyroxine (T4)
Description: Cmax was obtained from the concentration time curve. Cmax[aj] was the maximum serum concentration in pre dose corrected data where pre dose corrected data was obtained by subtracting pre dose level of Levothyroxine (T4) from level of Levothyroxine (T4) after administration.
Time Frame: Pre-dose, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.25, 3.5, 3.75, 4.0, 4.25, 4.5, 4.75, 5.0, 5.5, 6.0, 6.5, 8.0, 10.0, 12.0, 24.0, 36.0 and 48.0 hours post-dose
Population: Pharmacokinetic (PK) analysis set included all randomized participants who received study medication in both treatment periods. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Refernece Eutirox®: Participants received single oral dose of Reference Eutirox® 600 mcg (3 tablets of 200 mcg) in either Treatment Period 1 or 2 under fasting conditions.
- Test Eutirox®: Participants received single oral dose of Test Eutirox® 600 mcg (3 tablets of 200 mcg) in either Treatment Period 1 or 2 under fasting conditions.
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 38 | 38
nanogram per milliliter (ng/mL) | 67.24 (15.77) | 66.44 (15.77)
Statistical Analysis 1: Comparison: Refernece Eutirox® vs Test Eutirox®; Test type: Equivalence — Bio-equivalence Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; Geometric mean ratio = 98.53, 90% CI 2-sided [94.55 to 102.68]

2. Primary Outcome: Area Under Serum Concentration-Time Curve From Time Zero to The Last Sampling Time in Pre Dose Corrected Data (AUC0-t [aj]) of Levothyroxine (T4)
Description: AUC0-t was defined as area under the curve of the serum concentration as a function of time, from time 0 until the last sampling time by means of the trapezoidal rule. AUC0-t [aj] was the area under the serum concentration-time curve from time zero to the last sampling time in pre dose corrected data where pre dose corrected data was obtained by subtracting pre dose level of Levothyroxine (T4) from level of Levothyroxine (T4) after administration.
Time Frame: as for outcome 1
Population: PK analysis set included all randomized participants who received study medication in both treatment periods. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 38 | 38
nanogram*hour per milliliter (ng*hr/mL) | 1738.65 (438.93) | 1693.89 (389.50)
Statistical Analysis 1: Comparison: Refernece Eutirox® vs Test Eutirox®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 97.59, 90% CI 2-sided [91.34 to 104.26]

3. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of Levothyroxine (T4)
Description: Tmax was obtained directly from serum concentration-time curve.
Time Frame: as for outcome 1
Population: PK analysis set included all randomized participants who received study medication in both treatment periods.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 43 | 43
hour | 3.52 (1.19) | 3.50 (1.14)

4. Secondary Outcome: Elimination Half-Life (t1/2) of Levothyroxine (T4)
Description: t1/2 was the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by elimination constant.
Time Frame: as for outcome 1
Population: PK analysis set included all randomized participants who received study medication in both treatment periods.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 43 | 43
hour | 186.40 (96.26) | 189.10 (102.07)

5. Secondary Outcome: Area Under The Curve of the Serum Concentration as a Function of Time, From Time Zero to The Last Sampling Time (AUC0-t) of Levothyroxine (T4)
Description: Area under the serum concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ).
Time Frame: as for outcome 1
Population: PK analysis set included all randomized participants who received study medication in both treatment periods.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 43 | 43
ng*hour/mL | 5229.98 (562.73) | 5218.87 (587.42)
Statistical Analysis 1: Comparison: Refernece Eutirox® vs Test Eutirox®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 99.73, 90% CI 2-sided [98.45 to 101.03]

6. Secondary Outcome: Maximum Serum Concentration (Cmax) of Levothyroxine (T4)
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: PK analysis set included all randomized participants who received study medication in both treatment periods.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 43 | 43
ng/mL | 139.80 (16.16) | 139.17 (19.24)
Statistical Analysis 1: Comparison: Refernece Eutirox® vs Test Eutirox®; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 99.26, 90% CI 2-sided [97.70 to 100.85]

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination
Description: Physical examination included assessments of the general appearance, skin and mucosa, superficial lymph nodes, head and neck, chest, abdomen, musculoskeletal, and neurological systems. Number of participants with clinically significant abnormalities in physical examination findings were reported. Investigator decided clinical significance.
Time Frame: Baseline up to Day 37
Population: Safety analysis set included all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 44 | 44
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital sign assessment included blood pressure, pulse rate, body temperature and respiration. Number of participants with clinically significant abnormalities in vital signs were reported. Investigator decided clinical significance.
Time Frame: Baseline up to Day 37
Population: Safety analysis set included all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 44 | 44
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: The laboratory measurements included hematology, blood chemistry and urinalysis. Number of participants with clinically significant abnormalities in laboratory parameters were reported. Investigator decided clinical significance.
Time Frame: Baseline up to Day 37
Population: Safety analysis set included all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 44 | 44
Participants | 0 | 2

10. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG)
Description: The ECG recordings were obtained after 5 minutes of rest in a semi-supine position. ECG recordings included rhythm, ventricular rate, PR interval, QRS duration, QT and QTc intervals. Number of participants with clinically significant abnormalities in ECG were reported. Investigator decided clinical significance.
Time Frame: Baseline up to Day 37
Population: Safety analysis set included all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 44 | 44
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. Number of participants with adverse events were reported.
Time Frame: Baseline up to Day 51
Population: Safety analysis set included all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Refernece Eutirox® | Test Eutirox®
Number analyzed (Participants) | 44 | 44
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: Baseline up to Day 51
Groups:
- Reference Eutirox®: Participants received single oral dose of Reference Eutirox® 600 mcg (3 tablets of 200 mcg) in either Treatment Period 1 or 2 under fasting conditions.
Arm/Group | Reference Eutirox® | Test Eutirox®
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 4/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reference Eutirox® (N=44) | Test Eutirox® (N=44)
Dizziness (Nervous system disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Elevated Alanine Aminotransferase (Investigations) | 0 | 2
Elevated Aspartate Aminotransferase (Investigations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03979274/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT03979274/SAP_001.pdf